CLINICAL TRIAL: NCT03119363
Title: Treating Cancer-Related Fatigue Through Systematic Light Exposure
Brief Title: Treating Cancer-Related Fatigue Through Systematic Light Exposure (Light for Fatigue Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Hackensack Meridian Health (Other)
Responsible Party: Principal Investigator, William H. Redd, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 14-0937/14-1130
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma; Fatigue
Keywords: cancer-related fatigue; circadian rhythms; light therapy; systematic light exposure; cancer survivors; oncology; Multiple Myeloma; Hematopoietic stem cell transplantation; Autologous stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma; Fatigue; Neoplasms

STUDY DESIGN:
Intervention Model Description: Potentially eligible ASCT survivors will be identified by HSCT physicians and nurses at each medical center. A research assistant (RA) will be introduced to survivors who express an interest in the research. An RA will explain the study and consent those who are eligible. Once informed consent is obtained, an RA will conduct the screening interview (including the FACIT-Fatigue scale and a psychiatric and sleep disorder screening). An RA will review a checklist of inclusion and exclusion criteria. This information will also be verified by a review of participants' medical charts before participation begins. Eligible study participants will be randomly assigned condition using a block randomization table prepared by our statistician. Participants who do not meet eligibility criteria or who decline participation will be informed that they have completed their participation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Light (Experimental): The experimental systematic light exposure consists of exposure to light to reduce cancer-related fatigue. This group will self-administer 30 minutes of light from commercially available light glasses (AYO) each morning for 4 weeks. The AYO light glasses is a lightweight pair of glasses that emits light from LEDs at a distance of 15 millimeters (15mm, 0.015m) from the eye.
  Interventions: Device: AYO light glasses (Experimental)
- Comparison Light (Active Comparator): The active comparator condition consists of exposure to light to reduce cancer-related fatigue. This group will self-administer 30 minutes of light from commercially available light glasses each morning for 4 weeks.
  Interventions: Device: AYO light glasses (Comparator)

INTERVENTIONS:
Device: AYO light glasses (Experimental) — The AYO does not contain UV or infra-red light; the light spectrum begins at approximately 420nm. The circadian-effective AYO is programed at over 100 lux with 470nm frequency and irradiance of 250 qW/cm2, which is 100% intensity level. Irradiance over lux itself with AYO light glasses is believed to be more representative due to light frequency and proximity to the eye. Traditional Lightbox usual measure is Lux , AYO can be seen as comparable to 1,000 lux light box. The device is classified as a device that is safe for the eyes in accordance with the international standard IEC 62471 and is independently certified by TÜV Rheinland. AYO complies with the EU's CE marking (CE EMC EN 55014, EN 61000-4-3) as well as other national regulatory directives. AYO also complies with the United States of America's FCC marking (FCC Title 47, Chapter 1, Part 15, Class B FCC VOC: 47 CFR PART 15 OCT, 2016. CLASS B ANSI C 63.4: 2014) as well as other national marking regulatory directives.
  Arms: Experimental Light
Device: AYO light glasses (Comparator) — The comparison group will wear the same AYO glasses, but with a circadian ineffective (sham) light. The circadian-ineffective (sham) is programed at 1% intensity, therefore according to our calculation and checks it is below circadian threshold of 2 lux as specified.
  Arms: Comparison Light

SUMMARY:
Cancer related fatigue (CRF) is the most common cancer side effect and can severely interfere with activities of daily living long after completion of medical treatment. Pharmacologic agents to treat CRF have been studied but there is insufficient evidence to recommend their use. Non-pharmacological interventions for CRF have also been studied but are costly to implement and involve significant patient burden. This study investigates a novel low-cost/ low-burden intervention: systematic light exposure to treat CRF. Two hundred survivors of multiple myeloma and Diffuse Large B-cell Lymphoma between 1 month and 5 years post-autologous stem cell transplant (ASCT) will be recruited from three medical centers. The light will be administered by a small, personal light glasses daily for 4 weeks. Outcomes will be assessed at five separate time points, including baseline and follow-up. The study will specifically address recommendations made for interventions for CRF from the NCI Clinical Trials Planning meeting (JNCI, 2013).The proposed study will: 1) be the first large multisite study with a carefully delineated comparison condition to investigate the effects of light on CRF among ASCT survivors; 2) focus on a distinct, homogenous patient population; 3) include only survivors who experience clinical levels of CRF; and 4) address possible psychological and biological mechanisms. This study will have major public health relevance as it will determine if an easy-to-deliver, inexpensive, and low patient burden intervention effectively reduces CRF.

DETAILED DESCRIPTION:
The proposed multi-site randomized controlled trial (RCT) will investigate a novel intervention, systematic light exposure (sLE), to treat cancer-related fatigue (CRF) among Multiple Myeloma (MM) and Diffuse Large B-Cell Lymphoma (DLBCL) following autologous stem cell transplantation (ASCT). Cancer related fatigue (CRF) is persistent exhaustion related to cancer and/or its treatment. CRF is the most common cancer side effect and can severely interfere with activities of daily living long after completion of all medical treatment. Pharmacologic agents to treat CRF have been studied but there is insufficient evidence to recommend their use. Non-pharmacological interventions for CRF (including yoga, cognitive behavior therapy, hypnosis, and exercise) have also been studied; however, such interventions are costly to implement and involve significant patient burden. sLE is a low-cost, low- burden intervention that we have found to have beneficial effects for patients post-ASCT. The investigators initial randomized trial for CRF found that certain light exposure was associated with clinically significant reductions in fatigue (effect size d=0.98) More relevant to the proposed research is the preliminary investigation with sLE to treat CRF in MM and DLBCL which found that patients receiving certain sLE reported significantly less fatigue ( p=0.052). The proposed RCT will test the efficacy of sLE on CRF. It will also assess the effect of sLE on sleep, depressive symptoms, and both activity and cortisol circadian rhythms as these related processes have been hypothesized as possible mechanisms of

sLE's effects on CRF. Two hundred survivors of multiple myeloma and Diffuse Large B-cell Lymphoma between 1 month and 5 years post-autologous stem cell transplant (ASCT) will be recruited from two medical centers.

The light will be administered by light glasses for 4 weeks. Outcomes will be assessed at five separate time points including baseline and follow-ups.

The researchers' preliminary research has established the feasibility of this proposal. Moreover, in the preliminary research, 75% of participants completed the preliminary trial and data from the light box compliance meters showed that participants used the light boxes 80% of the days that treatment was scheduled. A large sample of fatigued MM and DLBCL ASCT survivors has been identified. The study will specifically address recommendations made for interventions for CRF from the NCI Clinical Trials Planning meeting (JNCI, 2013). It will: 1) be the first large multisite study with a carefully delineated comparison condition to investigate the effects of light on CRF among cancer survivors treated with ASCT; 2) focus on a distinct, homogenous patient population (MM and DLBCL ASCT survivors); 3) include only survivors who experience clinical levels of CRF; and 4) address possible mechanisms. This RCT will have major public health relevance as it will determine if an easy-to-deliver, inexpensive, and low patient burden intervention reduces CRF.

ELIGIBILITY:
Inclusion Criteria:

* In remission (partial to complete remission) verified by medical records
* With a history of ASCT as treatment for hematological malignancies such as MM, DLBCL, and related diseases and who are between one month and five years post-transplant

AND:

-With a score equal to or less than 33 on the FACIT-Fatigue scale (see below)

AND:

-Who are currently over age 18 and were at least age 16 at the time of ASCT

Exclusion Criteria:

* COVID diagnoses (active COVID-19) at the time of recruitment
* Under age 18
* Pregnancy
* Confounding underlying medical illnesses which may cause fatigue (e.g., severe Anemia not controlled by medication, per self-report corroborated by medical chart review (e.g., Hb<10gm/dl) )
* Severe sleep disorders (e.g. Narcolepsy)
* Eye Diseases which limit the ability of light to be processed (e.g., untreated cataracts, glaucoma that causes visual impairment, macular degeneration, blindness, pupil dilation problems or retina damage)
* Severe psychological impairment (e.g., hospitalization for depressive episode in the past 12 months)
* Currently employed in night shift work
* Previous use of light therapy to alleviate fatigue or depressive symptoms
* Self-reported history of bipolar disorder or manic episodes (which is a contra-indication for light treatment)
* Severe Psychiatric disorders assessed by the Psychoticism-Paranoia Screener
* Secondary cancer diagnosis (prior or current) within the past 5 years
* Plans to travel across meridians during the study

To decrease sample heterogeneity (consistent with JNCI, 2013 recommendations), allogeneic-HSCT survivors will not be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
FACIT-Fatigue Scale | 4 Years
  Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Scale. 13-item scale, each item 0=not at all to 4=very much, with higher score indicating more fatigue

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 4 years
  Sleep quality measured subjectively by the PSQI. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Rest/activity cycles | 4 years
  Sleep quality measured objectively by actigraphy. Actigraphy is a non-invasive method of monitoring rest/activity cycles.
Center for Epidemiologic Studies Depression Scale (CES-D) | 4 years
  Scoring for All Except Questions 4, 8, 12, and 16:
  * 0 points Rarely or none of the time (< 1 day)
  * 1 point Some or a little of the time (1-2 days)
  * 2 points Occasionally or a moderate amount of the time (3-4 days)
  * 3 points Most or all of the time (5-7 days)
  For questions 4, 8, 12, and 16, the scoring is exactly the same except that it is reversed: "Most or all of the time" is scored 0 points, "Rarely or none of the time" is scored 3 points Screening test score ranges are less than 15 = no depression, 15-21 = mild to moderate depression, and over 21 = possibility of major depression.
Correlation between sLE (or "Experimental Light") and depressive changes | 4 years
  Examine whether the effects of sLE on CRF are mediated by changes in depressive symptoms
Correlation between sLE (or "Experimental Light") and circadian rhythms | 4 years
  Examine whether the effects of sLE on CRF are mediated by changes in rest/activity circadian rhythms.
Correlation between Experimental Light compared with Comparison Light and cortisol circadian rhythm | 4 years
  Examine whether the Experimental Light compared with Comparison Light normalizes cortisol circadian rhythms and whether the effects of sLE on CRF are mediated by changes in cortisol circadian rhythms.
General Anxiety Disorder 7-item questionnaire (GAD-7) | 4 years
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire that asks user to rank how often they have been bothered by seven problems over the past two weeks from "0" (not at all) to "3" (nearly every day). The items that users are asked to rank levels of nervousness, anxiousness, relaxing, restlessness, irritability and fearfulness. Full scale from 0-21, with higher score indicating more symptoms.
Positive and Negative Affect Schedule (PANAS) | 4 years
  PANAS is a 20-item scale. Each item rated on a 5-point scale of 1 (not at all) to 5 (extremely), each subscale from 10-50, with higher score indicating more symptoms.
Patient Assessment of Own Functioning - PAOFI | 4 years
  Patient Assessment of Own Functioning - PAOFI is a 33-item instrument measuring four areas: memory, language and communication, motor/sensory-perceptual, higher level cognitive, and intellectual functions. Each item is rated from 0 (almost never) to 5 (almost always) for experiencing difficulty. Subscales: memory (0-45), language and communication (0-40), sensory-motor (0-25), intellectual (0-45), with total scale 0-155, with higher score indicating lower functioning
Multidimensional Fatigue Symptom Inventory - Short Form | 4 years
  Multidimensional Fatigue Symptom Inventory - Short Form is a 30-item scale, each item from 1 (not at all) to 4 (extremely), full scale from 24-95, with higher score indicating higher levels of fatigue
The Beck Depression Inventory II (BDI-II) | 4 years
  The Beck Depression Inventory II (BDI-II) is a 21 item self-report inventory measuring the severity of depression. Scoring is from 0 (minimal) to 3 (severe), with total score from 0-63. Higher total scores indicate more severe depressive symptoms.
Impact of Event Scale - Revised (IES-R) | 4 years
  Impact of Event Scale - Revised (IES-R) A 22-item self-report questionnaire measuring PTSD symptoms. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score ranging from 0 - 88 with higher score indicating more impact. Not a tool for diagnosis
Self Compassion Scale -SCS | 4 years
  Self Compassion Scale -SCS - 26-item instrument, full score from 1-5, with higher score indicating higher self compassion
Brief Symptom Inventory-18 (BSI-18) | 4 years
  Brief Symptom Inventory-18 (BSI-18) - self-report 18-item instrument. Scores on the 18 items are summarized on the Global Severity Index. Raw scores are converted to t-scores.
Posttraumatic Growth Inventory - (PTGI) Short Form | 4 years
  Posttraumatic Growth Inventory - (PTGI) Short Form - 10-item instrument, each item scored 0 (no change) to 5 (great degree change), full scale from 0-50, with higher score indicating greater growth.
Connor-Davidson Resilience Scale (CD-RISC-10) | 4 years
  The CD-RISC-10 is a 10 item ordinal scale rated on a 5-point scale: 0 (not true at all) to 4 (true nearly all the time). Full scale from 0-40, with higher scores reflecting greater resilience.
The Social Constraints Scale (SCS) | 4 years
  The Social Constraints Scale (SCS) - The SCS is a 15-item measure that reflects social conditions which cause a trauma survivor to feel unsupported, misunderstood, or otherwise alienated from their social network when they are seeking social support or attempting to express trauma-related thoughts, feelings, or concerns. Each item is scored 1 (never) to 4 (always). Full scale from 15-60, with higher score indicating the more often the person perceive they must inhibit themselves from expressing trauma-related thoughts and feelings to others.
C/E- Credibility/Expectancy Questionnaire | 4 years
  C/E- Credibility/Expectancy Questionnaire - A scale measuring treatment expectancy and rationale credibility for use in clinical outcome studies. Full scale from 0-10, with higher score indicating higher treatment expectancy
The Anxiety Sensitivity Index-3 - (ASI-3) | 4 years
  The Anxiety Sensitivity Index-3 - (ASI-3) is an 18 item measure, each item from 0 (very little) to 4 (very much), there are 3 subscales (physical, cognitive, and social) with each subscale range from 0-24 and the full scale range from 0 - 72, with higher scale indicating higher agreement.
MEQ- SA - Morningness Eveningness Questionnaire | 4 years
  MEQ- SA - Morningness Eveningness Questionnaire is a 19 item self-rated instrument to determine morningness-eveningness in human circadian rhythms. Full scale from 16-86, with higher score indicating the more the human circadian rhythm is of morning type.
Perceive Stress Scale (PSS) | 4 years
  Perceive Stress Scale (PSS) - A 10-item questionnaire, each item scored 0 (never) to 4 (very often), full scale from 0-40, with higher score indicating higher perceived stress.
Social Provision Scale | 4 years
  Social Provision Scale - 24 item instrument, each item scored (1) strongly disagree to (4) strongly agree. Full scale from 24 to 96, with higher score indicating higher perception of receiving provision.

CONTACTS AND LOCATIONS:
Overall Officials: William H Redd, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No